CLINICAL TRIAL: NCT06248255
Title: Impact to Skin Due to Wet Pad Application. Skin Status and Change in the Stratum Corneum as Measured With 4 Instruments in an Elderly Population.
Brief Title: Impact on Elderly Skin Due to Wet Pad Application.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DROPBOX
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Incontinence

STUDY DESIGN:
Intervention Model Description: The test pads is to both forearms of the participants. Participants will be blinded to the test pad type. In total 4 pads are applied per participant. The test pads are either Dry (control), 50% or at 100% capacity. Dry and 50% pads are applied once, 100% capacity twice. This to allow one pad for recovery measurement and one for water profile measurement. Pad location will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Single arm study, all participants get pads applied to their forearms
  Interventions: Other: Pads

INTERVENTIONS:
Other: Pads — Single arm design in which each participant act as its own control. Wet or Dry pads are applied to the participants forearms.

SUMMARY:
The clinical study aims to measure the changes in the stratum corneum on older healthy participants due to the application of a wet pad on the forearm. Participants are subject to baseline measures of TransEpidermalWaterLoss (TEWL), skin hydration (SH), pH and water profile (raman spectroscopy). Dry or wet pads are then added to the skin and worn for two hours. After a recovery period, the SkinSurfaceWaterLoss (SSWL) and skin hydration and water profile is measured. The study is conducted over a single visit. Pads on the arms consist of incontinence product cutouts and are loaded to 50% or 100% capacity. The endpoints are the changes in stratum corneum as measured by the instruments during the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 65 years.
2. Mentally and physically able to participate in this study.
3. Written informed consent to participate in this study.
4. Intact skin on the volar forearms without skin irritation.

Exclusion Criteria:

1. Have any known allergies or intolerances to one or several components of the absorbing incontinence product.
2. Suffer from excessive sweating, hyperhidrosis.
3. Have any other condition that makes participation in the clinical investigation inappropriate, as judged by investigator.
4. Not be of childbearing potential.
5. Have an alcohol and/or drug dependency.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change Trans Epidermal Water loss | 2 hours
  As measured by Dermalab instrument. Transepidermal water loss (TEWL) from dry skin and the subsequent skin surface water loss (SSWL) from wet skin
Change in skin hydration | 2 hours
  Skin hydration (SH) as measured with moisturemeter instrument
Change in Skin water profile | 2 hours
  As measured Confocal raman microspectometry. The water content of skin at different depths.

SECONDARY OUTCOMES:
Change in skin surface pH | 2 hours
  Skin surface pH measurement using pH meter

CONTACTS AND LOCATIONS:
Overall Officials: Shabira Abbas, PhD, Principal Investigator — Essity Hygiene and Health AB
Locations (1):
- Essity Study Site, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No